CLINICAL TRIAL: NCT06937450
Title: Traumatic Hemothorax Treatment With 14-Fr Pigtail Catheters or Large Bore (~28Fr) Chest Tubes With Daily Irrigation: A Pilot Single-Arm Intervention Study
Brief Title: Traumatic Hemothorax Drainage and Daily Lavage: Pilot Study
Acronym: HTXDLYLAVGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: CLR Medical (Unknown)
Responsible Party: Principal Investigator, Jeremy Cannon, Trauma Program Medical Director and Section Chief of Trauma, University of Pennsylvania
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 855480
Record Dates: First submitted 2024-03-21; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Hemothorax; Traumatic
MeSH Terms: conditions — Hemothorax | interventions — Drainage

STUDY DESIGN:
Intervention Model Description: This is a single arm interventional pilot study comparing groups of trauma hemothorax-diagnosed patients. There will be 2 treatment groups and 2 historical control groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Open 28 Fr Tube Thoracostomy with Daily Lavage and Drainage (Experimental): Open Tube Thoracostomy with Daily Lavage and Drainage
  Interventions: Device: CLR Irrigator; Procedure: Serial Lavage and Drainage; Device: 28 Fr Open Chest Tube
- Percutaneous 14-Fr Catheter with Daily Lavage and Drainage (Experimental): Percutaneous 14-Fr Catheter with Daily Lavage and Drainage
  Interventions: Device: CLR Irrigator; Procedure: Serial Lavage and Drainage; Device: Percutaneous 14Fr Chest Tube

INTERVENTIONS:
Device: CLR Irrigator — All enrolled patients will have their hemothorax treated with a CLR device that allows for easy suction and irrigation through indwelling catheters,
Procedure: Serial Lavage and Drainage — The current protocol is to do a singular lavage and drainage, this study will investigate the benefits of daily lavage.
Device: 28 Fr Open Chest Tube — Patients will have a standard 28 Fr open chest tube or a percutaneous 14Fr chest tube placed.
  Arms: Open 28 Fr Tube Thoracostomy with Daily Lavage and Drainage
Device: Percutaneous 14Fr Chest Tube — Patients will have a standard 28 Fr open chest tube, or a percutaneous 14Fr chest tube placed.
  Arms: Percutaneous 14-Fr Catheter with Daily Lavage and Drainage

SUMMARY:
This HTX treatment study evaluates the effects of chest tube size and the benefits of daily irrigations on acute HTX. 20 acutely injured but stable trauma patients requiring a chest tube for HTX will be enrolled. Patients will be assigned a 28Fr or 14 Fr chest tube with serial lavage and drainage. The endpoints will be HTX volume (by CT scan), complications, additional interventions, hospital length of stay, chest tube duration, provider feedback, and patient-reported outcomes.

DETAILED DESCRIPTION:
This hemothorax (HTX) treatment study will evaluate the effects of chest tube size and daily lavage on HTX management outcomes. A total of 20 stable trauma patients requiring a chest tube for HTX will be recruited and consented. These patients will then undergo either 28Fr or 14Fr chest tube placement, depending on the preference of the treatment team at the time of placement. The study will include 10 patients with each type of chest tube (28Fr and 14Fr). Daily lavage will then be performed at 24h and 48h post-placement. Patients will be compared to historical control patients from the trauma registry who received either 28Fr or 14Fr chest tube placement followed by an initial lavage only. The primary endpoint will be the need for additional interventions such as tPA, additional chest tubes, thoracoscopic surgery (VATS), or thoracotomy. Secondary endpoints will include X-ray appearance at 72 hours, volume of HTX on CT at 72 hours, procedural complications, development of empyema (safety endpoint), development of delayed bleeding (safety endpoint), hospital length of stay, chest tube duration, provider feedback, and patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide consent for the research study
2. More than 15 years of age
3. Presence of acute traumatic HTX or HTX-PTX diagnosed on chest CT scan within 24 hours of injury and clinical indication for drainage (hemothorax of moderate or large size greater then 300 mL)
4. Hemodynamic stability (heart rate 120 beats per minute; systolic blood pressure 90 mmHg)
5. Bilateral or unilateral hemothorax of greater than 300 mL HTX by Mergo Formula from chest CT
6. Able to complete the entire study including randomization, tube placement, lavages and final CT Scan.

Exclusion Criteria:

1. Less than 15 years of Age
2. Prisoner
3. Pregnant due to the risk of CT scans
4. HTX or HTX-PTX not requiring drainage or drainage performed prior to randomization/enrollment
5. Patients undergoing operative intervention (i.e. thoracotomy) as initial management of hemothorax (6) Persistent hemodynamic instability after initial resuscitation and CT imaging

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Remaining Hemothorax Volume at 72 hours | 72 hours
  Assessed by CT and Mergo Formula

SECONDARY OUTCOMES:
Number of patients requiring intervention for retained hemothorax (excluding those who require intervention for other treatment) | Through hospital discharge or 30 days
  All interventions focused on resolving any remaining hemothorax
Patient Tolerability - Numerical Rating Scale (NRS) Perception Experience (IPE) | 1 hour, 24 hours, 48 hours
  Patient perception of the drainage and lavage procedure. Did this Drainage and Lavage procedure resolve, lessen or worsen the patient's symptoms?
Patient Tolerability - Insertion Perception Experience (IPE) Perception Experience (IPE) | 1 hour
  Patient perception of the chest tube insertion procedure.
  1. = It was okay, I can tolerate it, I can do it again.
  2. = It was okay, but I don't want to go through this again.
  3. = It was a bad experience for me.
  4. = It was a worse experience for me.
  5. = It was the worst experience of my life!
Ease of CLR System Use - Industry-Standard System Usability Scale (SUS) | 1 hour, 24 hours, 48 hours
  By physician who used the CLR Irrigator System. 5-point Likert scale from strongly disagree (low) to strongly agree (high).
Chest Tube Placement Duration | Through discharge or 30 days
  Length of time the chest tube remained in the patient
Length of hospital stay | Through discharge or 30 days
  Length of hospital stay
Aggregate Hospital Charges for Patient Stay | Through discharge or 30 days
  Estimated cost of patient care at hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Cannon, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share Individual Participant Data.